CLINICAL TRIAL: NCT04824911
Title: Early Intensive Medical Therapy for the Prevention of Early Neurological Deterioration in Branch Atheromatous Disease
Brief Title: Statin and Dual Antiplatelet Therapy to Prevent Early Neurological Deterioration in Branch Atheromatous Disease
Acronym: SATBRAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202001386A3
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acute Stroke; Dual Antiplatelet Therapy; Statin
Keywords: Branch Atheromatous Disease; Early neurological deterioration; Dual antiplatelet therapy; Statin
MeSH Terms: conditions — Stroke | interventions — Clopidogrel; Aspirin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This group will receive dual antiplatelet and high-intensity statin treatment.
  * Dual antiplatelet treatment: loading of clopidogrel 300mg plus aspirin 300mg, followed by clopidogrel 75 mg/day and aspirin 100 mg/d from day 2 to day 21, and followed by clopidogrel 75 mg/d or aspirin 100 mg/d from day 15 to day 90.
  * High-intensity statin treatment: Atorvastatin 40-80mg/day or Rosuvastatin 20 mg/day for 90 days.
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: Atorvastatin; Drug: Rosuvastatin
- Historical control (Active Comparator): A historical control group of patients receiving single antiplatelet therapy but no high-intensity statin treatment will be drawn from previous prospective observation studies. Antiplatelet therapy includes aspirin(100-300mg/day) or Clopidopgrel (75mg/day).
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — 300mg loading and 75mg/day from day 2
Drug: Aspirin — Aspirin(100-300mg/day)
Drug: Atorvastatin — Atorvastatin 40-80mg/day
  Arms: Intervention group
Drug: Rosuvastatin — Rosuvastatin 20 mg/day.
  Arms: Intervention group

SUMMARY:
Branch atheromatous disease (BAD) has been reported to contribute to small-vessel occlusion and is associated with a higher possibility of early neurological deterioration (END). Because the pathology of BAD is due to atherosclerosis, the investigators postulate that early intensive medical treatment with dual antiplatelet therapy(DAPT) and high-intensity statin may prevent END and recurrent stroke. The investigators hypothesise that intensive medical therapy can prevent END in BAD using aspirin, clopidogrel and high-intensity statin.

DETAILED DESCRIPTION:
The SATBRAD study is a single-centre, prospective, open-label, single-group trial with a historical control group of BAD patients treated with single antiplatelet therapy and regular statin treatment in Chang Gung Memorial Hospital in Taiwan.

Eligible participants are as follows:

1. have a clinical diagnosis of ischemic stroke;
2. National Institute of Health Stroke Scale (NIHSS) score of 1-8;
3. an ischemic lesion on diffuse-weighted imaging located in the middle cerebral artery(MCA) perforator, Heubner's artery or vertebrobasilar perforator territories;
4. BAD, defined by a visible lesion in three or more axial MRI cuts in the MCA perforator territory or Heubner's artery territories or infarcts that extended from the basal surface of the brainstem.
5. can receive intensive medical treatment within 24 hours of stroke onset.

Participants in the intervention group will receive DAPT and high-intensity statin treatment. DAPT treatment is administered within 24 hours of stroke onset, with aspirin (300 mg loading and 100 mg/day) and clopidogrel (300mg and 75m/day). Participants will take aspirin and clopidogrel for 21 days and then keep aspirin or clopidogrel alone. High-intensity statin is administered, including atorvastatin 40-80mg or rosuvastatin 20 mg for 3 months.

A historical control group of patients receiving single oral antiplatelet medication and regular statin treatment will be drawn from previous prospective observation studies which were executed since Jan. 2011 to Dec. 2020. The total sample sizes are 147 for intervention group and 277 for control group.

The primary endpoint is the composite of END, defined as an increase of ≧2 points of NIHSS within 7 days, and recurrent ischemic stroke within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke with National Institute of Health Stroke Scale (NIHSS) score of 1-8
* An ischemic lesion on diffuse-weighted imaging located in the MCA perforator, or Heubner's artery territories or vertebro-basilar perforator territories at brain stem.
* Branch atheromatous disease, defined by a visible lesion in three or more axial MRI cuts in the MCA perforator or Heubner's artery territories or infarcts that extended from the basal surface of the brainstem.
* Ability to randomize within 24 hours of time last known free of new ischemic symptoms.
* Head CT or MRI ruling out hemorrhage or other pathology, such as vascular malformation, tumor, or abscess, that could explain symptoms or contraindicate therapy.
* Ability to tolerate high intensity medical therapy, including aspirin at a dose of 50-325 mg/day, clopidogrel with 300mg loading and 75mg after day 2 and high-intensity statin(either atorvastatin 40-80mg or rosuvastatin 20 mg/day).
* Pre-stroke mRS≦1

Exclusion Criteria:

* Age < 20 years.
* In the judgment of the treating physician
* A candidate for thrombolysis, endarterectomy or endovascular intervention.
* Receipt of any intravenous or intra-arterial thrombolysis within 1 week prior to index event.
* Patients with more than 50% stenosis of the relevant arteries on magnetic resonance angiography (MRA), including intra- or extra-cranial internal carotid artery, middle cerebral artery or basilar artery.
* Patients with high risk of cardioembolic source, such as atrial fibrillation, acute myocardial infarction, severe heart failure or valvular heart disease.
* Other determined stroke etiology, such as vasculitis, shock, antiphospholipid antibody syndrome and etc.
* Gastrointestinal bleed or major surgery within 3 months prior to index event.
* History of nontraumatic intracranial hemorrhage.
* Clear indication for anticoagulation during the study period (deep venous thrombosis, pulmonary embolism or hypercoagulable state).
* Qualifying ischemic event induced by angiography or surgery.
* Severe non-cardiovascular comorbidity with life expectancy <3 months.
* Contraindication to clopidogrel, aspirin, atorvastatin or rosuvastatin
* Known allergy to clopidogrel, aspirin atorvastatin or rosuvastatin
* Severe renal (serum creatinine >2 mg/dL) or hepatic insufficiency (INR>1.2; ALT>40 U/L or any resultant complication, such as variceal bleeding, encephalopathy, or jaundice)
* Hemostatic disorder or systemic bleeding in the past 3 months
* Current thrombocytopenia (platelet count <100 x109/L) or leukopenia (<2 x109/L)
* History of drug-induced hematologic or hepatic abnormalities
* Anticipated requirement for long-term (>7 day) non-study antiplatelet drugs (e.g., dipyridamole, ticagrelor, ticlopidine), or NSAIDs.
* Low-density lipoprotein<70mg/dl without prior statin treatment in recent one year or within 2 days after recruitment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with early neurological deterioration within 7 days and recurrent ischemic stroke within 30 days. | 30 days
  The early neurological deterioration is defined as an increase of 2 points of NIHSS.
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The maximum possible score is 42, with the minimum score being a 0.

SECONDARY OUTCOMES:
Percentage of patients with favorable functional recovery defined as a mRS ≦1 | 90 days
  Defined as a mRS ≦1. The Modified Rankin Scale (mRS) runs from 0-6, running from perfect health without symptoms(score 0) to death(score 6).
Percentage of patients with new clinical vascular events | 90 days
  ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death
Changes of atherosclerotic plaque | 6 months
  The changes of atherosclerotic plaque was measured by high-resolution MRI initially and 6 months later.
Numbers of moderate to severe bleeding events | 90 days
Total mortality | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Yenchu Huang, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charidimou A, Pantoni L, Love S. The concept of sporadic cerebral small vessel disease: A road map on key definitions and current concepts. Int J Stroke. 2016 Jan;11(1):6-18. doi: 10.1177/1747493015607485. PMID 26763016
- [Background] Petrone L, Nannoni S, Del Bene A, Palumbo V, Inzitari D. Branch Atheromatous Disease: A Clinically Meaningful, Yet Unproven Concept. Cerebrovasc Dis. 2016;41(1-2):87-95. doi: 10.1159/000442577. Epub 2015 Dec 16. PMID 26671513
- [Background] Yamamoto Y, Ohara T, Hamanaka M, Hosomi A, Tamura A, Akiguchi I. Characteristics of intracranial branch atheromatous disease and its association with progressive motor deficits. J Neurol Sci. 2011 May 15;304(1-2):78-82. doi: 10.1016/j.jns.2011.02.006. Epub 2011 Mar 13. PMID 21402390
- [Background] Kim JS, Yoon Y. Single subcortical infarction associated with parental arterial disease: important yet neglected sub-type of atherothrombotic stroke. Int J Stroke. 2013 Apr;8(3):197-203. doi: 10.1111/j.1747-4949.2012.00816.x. Epub 2012 May 9. PMID 22568537
- [Background] Gao S, Wang YJ, Xu AD, Li YS, Wang DZ. Chinese ischemic stroke subclassification. Front Neurol. 2011 Feb 15;2:6. doi: 10.3389/fneur.2011.00006. eCollection 2011. PMID 21427797
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Kimura T, Tucker A, Sugimura T, Seki T, Fukuda S, Takeuchi S, Miyata S, Fujita T, Hashizume A, Izumi N, Kawasaki K, Katsuno M, Hashimoto M, Sako K. Ultra-Early Combination Antiplatelet Therapy with Cilostazol for the Prevention of Branch Atheromatous Disease: A Multicenter Prospective Study. Cerebrovasc Dis Extra. 2016;6(3):84-95. doi: 10.1159/000450835. Epub 2016 Oct 12. PMID 27728903
- [Background] Wang C, Yi X, Zhang B, Liao D, Lin J, Chi L. Clopidogrel plus aspirin prevents early neurologic deterioration and improves 6-month outcome in patients with acute large artery atherosclerosis stroke. Clin Appl Thromb Hemost. 2015 Jul;21(5):453-61. doi: 10.1177/1076029614551823. Epub 2014 Sep 23. PMID 25248816
- [Background] Kim D, Park JM, Kang K, Cho YJ, Hong KS, Lee KB, Park TH, Lee SJ, Kim JG, Han MK, Kim BJ, Lee J, Cha JK, Kim DH, Nah HW, Kim DE, Ryu WS, Kim JT, Choi KH, Choi JC, Lee BC, Yu KH, Oh MS, Kim WJ, Kwon JH, Shin DI, Sohn SI, Hong JH, Lee JS, Lee J, Gorelick PB, Bae HJ. Dual Versus Mono Antiplatelet Therapy in Large Atherosclerotic Stroke. Stroke. 2019 May;50(5):1184-1192. doi: 10.1161/STROKEAHA.119.024786. PMID 30932785
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Fang JX, Wang EQ, Wang W, Liu Y, Cheng G. The efficacy and safety of high-dose statins in acute phase of ischemic stroke and transient ischemic attack: a systematic review. Intern Emerg Med. 2017 Aug;12(5):679-687. doi: 10.1007/s11739-017-1650-8. Epub 2017 Mar 16. PMID 28303440
- [Background] Chung JW, Cha J, Lee MJ, Yu IW, Park MS, Seo WK, Kim ST, Bang OY. Intensive Statin Treatment in Acute Ischaemic Stroke Patients with Intracranial Atherosclerosis: a High-Resolution Magnetic Resonance Imaging study (STAMINA-MRI Study). J Neurol Neurosurg Psychiatry. 2020 Feb;91(2):204-211. doi: 10.1136/jnnp-2019-320893. Epub 2019 Aug 1. PMID 31371644
- [Background] Siegler JE, Martin-Schild S. Early Neurological Deterioration (END) after stroke: the END depends on the definition. Int J Stroke. 2011 Jun;6(3):211-2. doi: 10.1111/j.1747-4949.2011.00596.x. PMID 21557807
- [Derived] Huang YC, Weng HH, Tsai YH, Lin LC, Lee JD, Yang JT, Pan YT. Early intensive therapy for preventing neurological deterioration in branch atheromatous disease. Ther Adv Neurol Disord. 2025 Jul 24;18:17562864251357274. doi: 10.1177/17562864251357274. eCollection 2025. PMID 40726739
- [Derived] Huang YC, Tsai YH, Lin LC, Weng HH, Lee JD, Yang JT. Preliminary results on temporal evolution and clinical implications of atherosclerotic plaque in branch atheromatous disease after statin treatment. Ther Adv Neurol Disord. 2024 Sep 18;17:17562864241273902. doi: 10.1177/17562864241273902. eCollection 2024. PMID 39314261
- [Derived] Huang YC, Lee JD, Weng HH, Lin LC, Tsai YH, Yang JT. Statin and dual antiplatelet therapy for the prevention of early neurological deterioration and recurrent stroke in branch atheromatous disease: a protocol for a prospective single-arm study using a historical control for comparison. BMJ Open. 2021 Nov 26;11(11):e054381. doi: 10.1136/bmjopen-2021-054381. PMID 34836908